CLINICAL TRIAL: NCT05546801
Title: Antenatal Ultrasound Diagnosis of Periventricular Pseudocysts and Postnatal Outcome
Acronym: UDiPPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2022/14
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Periventricular Pseudocysts
Keywords: periventricular pseudocysts; postnatal development
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: questionnaire on postnatal development
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- questionnaire (Experimental): Questionnaire on postnatal development
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaire on postnatal development

SUMMARY:
The present study aims to improve the information given to the parents during the screening of periventricular pseudocysts in the Pluridisciplinary Center of Prenatal Diagnosis, with retrospective cases screened during the last 5 years in university hospital of Bordeaux.

DETAILED DESCRIPTION:
Antenatal ultrasound screening for periventricular pseudocysts is steadily increasing, enabled in part by technological advances in ultrasound equipment.

Most of studies dealing with periventricular pseudocysts and subsequent neurodevelopment are based on neonatal screening, mostly performed in neonatal units.

Current data in the literature on the postnatal outcome of children screened antenatally are scarce; there are only 5 cohort studies with small numbers on the subject.

The present study aims to improve the information given to the parents during the screening of periventricular pseudocysts in the Pluridisciplinary Center of Prenatal Diagnosis, with retrospective cases screened during the last 5 years in university hospital of Bordeaux.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient diagnosed with a periventricular cyst during a prenatal ultrasound at Bordeaux University Hospital between January 1, 2016 and December 31, 2020.
* Patient affiliated with or benefiting from a social security plan.
* Oral informed consent.

Exclusion Criteria:

* Subarachnoid cyst
* Blake's pouch cyst
* Choroid plexus cyst
* Periventricular leukomalacia
* Poor understanding of French
* Patient under legal protection.

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
postnatal child development | Baseline
  composite criterion as follows: Delayed acquisition is defined according to the standards of the Pediatric Society: age of sitting > 8 months, age of walking > 18 months, ability or not to associate 3 words at age 3. The use of a medical profession concerns follow-up by a speech therapist, a psychomotrician or a physiotherapist. It is not necessarily a periodic follow-up but a minimum of 2 consultations after the "assessment" consultation.
  The scoring defines 2 groups,
  * children with 0 points considered with a "normal" post-natal development
  * children with 1 point or more considered with a post-natal development disorder.

SECONDARY OUTCOMES:
mother's medical history | Baseline
  mother's medical history
medical history of the child | Baseline
  medical history of the child

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No